CLINICAL TRIAL: NCT05264298
Title: Video-based Intervention to Reduce Treatment and OUtcome Disparities in Adults Living With Stroke or Transient Ischemic Attack (VIRTUAL)
Brief Title: Video-based Intervention to Address Disparities in Blood Pressure Control After Stroke
Acronym: VIRTUAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Anjail Z Sharrief, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSC-MS-21-0549; 1R01MD016465-01 (NIH)
Record Dates: First submitted 2022-02-06; First posted 2022-03-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VIRTUAL Intervention (Treatment) (Experimental): Participants assigned to intervention arm will have scheduled video telehealth appointments with a multidisciplinary team (Stroke provider, social worker, pharmacist) and remote telemonitoring of blood pressure with blood pressure medication adjustments biweekly as needed by pharmacists.
  Interventions: Other: VIRTUAL
- Standard Care (Active Comparator): Participants assigned to standard care will follow-up with a stroke provider within 2 weeks of discharge and primary care as per usual recommendations. Participants will monitor their blood pressure on their own and pharmacists will contact participants monthly to review blood pressure. Pharmacists will make recommendations for blood pressure medication adjustment to participant primary care provider.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: VIRTUAL — At the time of discharge, stroke survivors in the VIRTUAL arm will receive a package containing an iPad and a remote BP monitoring device that allows transmission of BP to the study team.The first telehealth visit will occur 7-14 days after discharge. Patient will be counseled on the importance of BP monitoring, salt reduction, and the importance of diet and exercise for stroke prevention. Medications, side effects and interactions will be reviewed. The social worker will refer the patient to specific resources according to social needs abd patient will be referred to a primary care provider if they do not have one. Subsequent video visits will be 1-month (30 days +/- 7) , 3 months (90 days +/- 14), and 5 months (150 days +/- 14) days after enrollment.
  Arms: VIRTUAL Intervention (Treatment)
Other: Standard care — Participants randomized to standard care will receive an educational packet and a blood pressure monitor prior to hospital discharge. They will be contacted by a social worker to determine if they received their medications and appointments. The stroke practitioner will evaluate the patients at 7-14 days and then follow up according to current standard of care. They will be seen over video or in-person, according to their preference and capabilities. The pharmacist will contact patients at 1-month (30 +/- 7 days) days over the telephone to review BP logs and will make recommendations to their primary care provider to adjust BP medications. Subsequent pharmacist calls will occur monthly until 6 months and recommendations for medication adjustments will be communicated to their primary care provider.
  Arms: Standard Care

SUMMARY:
The purpose of this study is to examine the impact of a multidisciplinary telehealth-based model of outpatient stroke care on blood pressure control following stroke, and further, to evaluate its impact on racial disparities in post-stroke blood pressure control.

DETAILED DESCRIPTION:
Blood pressure is poorly controlled for many stroke survivors and racial disparities in blood pressure control and stroke recurrence exist.

The purpose of this study is to examine the impact of a multidisciplinary, telehealth based, outpatient model of care on outcomes after stroke with a focus on blood pressure control. The Video-based Intervention to Reduce Treatment and Outcome Disparities in Adults Livings with Stroke and Transient Ischemic Attack (VIRTUAL) has several components including early follow-up via telehealth with a multidisciplinary team, remote blood pressure monitoring, and medication adjustment by a pharmacist.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke, hemorrhagic stroke (intracerebral hemorrhage),or transient ischemic attack (TIA
* Presence of hypertension (by clinical history or hospital BP ≥140/90 mmHg on two occasions)
* Plan to discharge home after stroke
* Ability to provide consent (patient or caregiver) in English or Spanish. Patients with cognitive impairment or aphasia limiting participation will be included if they have a caregiver to assist with monitoring and telehealth visits.
* Two neurologists must agree on TIA diagnosis

Exclusion Criteria:

* Modified Rankin scale (mRs) > 4 (severe disability) at time of discharge
* Life expectancy < 1 year or terminal illness
* Stroke unrelated to vascular risk factors (RFs) (drug use, trauma, vasculitis)
* Pregnancy
* Symptomatic flow limiting carotid stenosis without plan for intervention
* Long-term BP goal ≥ 130/80 mmHg according to clinical team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
6 month blood pressure control (24-hour ambulatory) | 6 months after discharge
  Proportion of participants with controlled BP according to 24- hour ambulatory BP (<125/75 mmHg)

SECONDARY OUTCOMES:
12 month blood pressure control (24-hour ambulatory) | 12 months after discharge
  Proportion of participants with controlled BP according to 24- hour ambulatory BP (<125/75 mmHg)
Composite Recurrent Vascular Events | 12 months after discharge
  Number of patients with myocardial infarction, ischemic or hemorrhagic stroke, coronary revascularization, acute cardiac death, and heart failure hospitalization)
Proportion of uninsured who obtain insurance | 3 months after hospital discharge
  Proportion of uninsured patients who obtain insurance
Proportion of uninsured who obtain insurance | 6 months after hospital discharge
  Proportion of uninsured patients who obtain insurance
Acute healthcare utilization | 3 months after hospital discharge
  Number of hospital readmissions, emergency department (ED) visits, and urgent care visits
Acute healthcare utilization | 6 months after hospital discharge
  Number of hospital readmissions, ED visits, and urgent care visits
Acute healthcare utilization | 12 months after hospital discharge
  Number of hospital readmissions, ED visits, and urgent care visits

OTHER OUTCOMES:
24 hour ambulatory systolic blood pressure | 6 month
  24 hour systolic blood pressure as assessed by an ambulatory blood pressure monitor
24 hour ambulatory systolic blood pressure | 12 month
  24 hour systolic blood pressure as assessed by an ambulatory blood pressure monitor
24 hour ambulatory diastolic blood pressure | 6 month
  24 hour diastolic blood pressure as assessed by an ambulatory blood pressure monitor
24 hour ambulatory diastolic blood pressure | 12 month
  24 hour diastolic blood pressure as assessed by an ambulatory blood pressure monitor
Daytime ambulatory systolic blood pressure | 6 month
  Daytime systolic blood pressure as assessed by an ambulatory blood pressure monitor
Daytime ambulatory systolic blood pressure | 12 month
  Daytime systolic blood pressure as assessed by an ambulatory blood pressure monitor
Daytime ambulatory diastolic blood pressure | 6 month
  Daytime diastolic blood pressure as assessed by an ambulatory blood pressure monitor
Daytime ambulatory diastolic blood pressure | 12 month
  Daytime diastolic blood pressure as assessed by an ambulatory blood pressure monitor
Night time ambulatory systolic blood pressure | 6 month
  Night time systolic blood pressure as assessed by an ambulatory blood pressure monitor
Night time ambulatory systolic blood pressure | 12 month
  Night time systolic blood pressure as assessed by an ambulatory blood pressure monitor
Night time ambulatory diastolic blood pressure | 6 month
  Night time diastolic blood pressure as assessed by an ambulatory blood pressure monitor
Night time ambulatory diastolic blood pressure | 12 month
  Night time diastolic blood pressure as assessed by an ambulatory blood pressure monitor
Proportion of participants who quit smoking or attempt to quit smoking | 6 months
  Among participants who are tobacco users at time of enrollment
Proportion of participants who quit smoking or attempt to quit smoking | 12 months
  Among participants who are tobacco users at time of enrollment
Proportion of participants who quit smoking | 6 months
  Among participants who are tobacco users at time of enrollment
Proportion of participants who quit smoking | 12 months
  Among participants who are tobacco users at time of enrollment
Depressive symptoms as assessed by score on the Patient Health Questionnaire 9 | 6 months
  Patient Health Questionnaire 9 total score ranges from 0 to 27
Depressive symptoms as assessed by score on the Patient Health Questionnaire 9 | 12 months
  Patient Health Questionnaire 9 total score ranges from 0 to 27

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Z Sharrief, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okpala M, Izeogu C, Wang M, Green C, Cooksey G, Nguyen T, Cohen S, Bryant L, Hernandez DC, Bernstam EV, Gonzales M, Conyers R, Chiadika O, Varacalli K, Savitz SI, Yamal JM, Sharrief AZ. Video-based Intervention to Reduce Treatment and Outcome Disparities in Adults Living with Stroke or Transient Ischemic Attack (VIRTUAL): protocol for a randomized controlled trial. Trials. 2025 Aug 12;26(1):288. doi: 10.1186/s13063-025-09003-5. PMID 40796883